CLINICAL TRIAL: NCT03318588
Title: Intravitreous CytokinE Level in pAtient With retiNal Detachment
Acronym: ICELAND
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Docteur Jean-Baptiste CONART, Medical Doctor, Central Hospital, Nancy, France
Other Study IDs: 2017-A02195-48
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Retinal Detachment
Keywords: Retinal detachment; Photoreceptor apoptosis; Cytokine
MeSH Terms: conditions — Retinal Detachment | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients undergoing vitrectomy for primary retinal detachment
  Interventions: Procedure: Vitrectomy
- Control: Patients undergoing vitrectomy for idiopathic macular hole
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy — Pars plana vitrectomy

SUMMARY:
Photoreceptor apoptosis is the basis for permanent visual loss in a number of retinal disorders including age-related macular degeneration (AMD) and retinal detachment (RD). Thus, despite tremendous advances in vitreoretinal surgery and management of rhegmatogenous RD leading to a primary reattachment rate over 95%, some patients show poor visual recovery because of photoreceptor apoptosis.

Physiologically, microglial cells (resident macrophages) are present only in the inner retina. The subretinal space, located between the retinal pigment epithelium (RPE) and the photoreceptor outer segments (POS), is devoid of all mononuclear phagocytes and form a zone of immune privilege. In AMD, several studies showed a strong association between subretinal mononuclear phagocytes infiltration and advanced forms of AMD. Experimental work in mice suggest that this infiltration plays an important role in the pathogenesis of this condition by producing inflammatory cytokines.

RD-induced photoreceptor apoptosis might result from similar mechanisms. The aim of this study is to determine the cytokine profile in vitreous samples from patients with RD and to compare it with those from control patients with macular hole.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary retinal detachment requiring vitrectomy
* Patients with idiopathic macular hole requiring vitrectomy

Exclusion Criteria:

* History of retinal detachment or intraocular inflammatory diseases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from the department of Ophthalmology (Nancy University Hospital)
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Intravitreous cytokine levels | up to one month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste CONART, MD, Principal Investigator — Brabois Hospital, Department of Ophthalmology
Locations (1):
- Brabois Hospital, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Conart JB, Blot G, Augustin S, Millet-Puel G, Roubeix C, Beguier F, Charles-Messance H, Touhami S, Sahel JA, Berrod JP, Leveillard T, Guillonneau X, Delarasse C, Sennlaub F. Insulin inhibits inflammation-induced cone death in retinal detachment. J Neuroinflammation. 2020 Nov 26;17(1):358. doi: 10.1186/s12974-020-02039-1. PMID 33243251